CLINICAL TRIAL: NCT01531582
Title: The Efficacy of Minocycline in the Treatment of Angelman Syndrome
Brief Title: Minocycline in the Treatment of Angelman Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WEEBER001
Record Dates: First submitted 2012-02-05; First posted 2012-02-13 (Estimated); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2015-11

CONDITIONS: Angelman Syndrome
Keywords: Angelman; Minocycline; cognitive; children; tetracycline
MeSH Terms: conditions — Angelman Syndrome; cyclopia sequence | interventions — Minocycline; Tetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Children with Angelman Syndrome (Experimental): Children with a molecularly confirmed diagnosis of Angelman Syndrome meeting the protocol requirements will be selected randomly. All participants will receive the study drug, minocycline, over an identical time course. Participants will undergo identical baseline, 8 and 16 week follow up assessments.
  Interventions: Drug: minocycline

INTERVENTIONS:
Drug: minocycline — The participant's parent or guardian will be instructed to administer minocycline caplets by mouth twice daily. Parents or guardians will be instructed to avoid dairy products, antacids, or any vitamin preparation that contains any divalent or trivalent cations (e.g. Aluminum, Calcium, Magnesium, etc.) for one hour prior to, and two hours after study medication administration.
  Other Names: Alti-Minocycline; Apo-Minocycline; Arestin; Dynacin; Gen-Minocycline; Klinomycin; Minociclina [INN-Spanish]; Minocin; Minocyclin; Minocycline HCl; Minocyclinum [INN-Latin]; Minocyn; Minomycin; Novo-Minocycline; Solodyn; Vectrin; Tetracycline

SUMMARY:
There is mounting evidence to suggest that a treatment for Angelman syndrome is not just possible, but probable. The lack of known molecular targets associated with AS has hampered the development of specific therapeutics. However, a recent surge of potential therapeutics for other disorders associated with cognitive disruption has begun to be used in human clinical trials. The molecular modes of action for many of these new therapeutic agents have correlates to counter the molecular defects observed in AS. One such agent is minocycline (MC), a drug traditionally used as an antibiotic. This compound administered to a mouse model of AS showed a significant decrease in motor deficit and an increase in long term potentiation. The investigators believe a similar result will be observed when minocycline is administered to the AS patient and may lead to the development of an effective AS therapeutic.

DETAILED DESCRIPTION:
This prospective single arm cohort study is to be conducted at the University of South Florida. The study will examine the effect minocycline (MC) has on the traits of Angelman Syndrome.

Minocycline HCl is an FDA approved antimicrobial medication in the tetracycline family of drugs. Of all the tetracyclines, MC is the most lipid soluble and most active. Unlike other antibiotics in this family, MC possesses the unique characteristic of being able to cross the blood brain barrier. The study dosage has been used in other trial treatments of other neurologic disorders with positive outcomes. Studies of long-term administration of MC at the study dose have been shown to be safe and well tolerated. This dosage has already been approved by the FDA for use in the treatment of bacterial infections of multiple organ systems, and acne vulgaris.

It is important to note that minocycline is not approved to treat Angelman syndrome or to be used in children younger than 8 years old. The study protocol has been reviewed by several physicians and scientists and been deemed safe to proceed. As with any medication the potential for side effects exist. The side effects range from serious to mild and include allergic reactions to upset stomach. In order to minimize this risk, the medical staff will perform a thorough medical history and physical examination before the prescription is issued to ensure no allergy to this medication, penicillin or another tetracycline exists. Discoloration of the teeth is potential adverse effect that exists when taking high doses of MC over long periods of time. The tooth discoloration is permanent and the parent or guardian of the participants will be made aware of this potential side effect prior to enrollment in the study. In other studies using MC, the most common complaint was gastrointestinal upset.

Recruitment & Prescreening - We anticipate some of the study participants will live far from the study site. In order to reduce screen failures (travel to the site only to find out your child doesn't meet the study criteria) the following process is required. To give parents the opportunity to consider the study and have time to consult with their doctor(s), we will begin recruitment approximately one week after the study has been published on this website. Parents will be asked to submit their information electronically by clicking the link at the bottom of this webpage or by accessing weeberlab.com/clinical_trials.html. In the event they do not have internet access, they may call the study coordinator for assistance. Once you have indicated your interest in participation, a packet of information will be sent to you via email (or postal service if you prefer). The packet will include an informed consent document, a release of medical information and a form for your primary care doctor to complete and return directly to us. All of this information will be reviewed by the medical staff to determine your child's eligibility. Out of the first 50 eligible participants, 24 will be randomly selected by the Clinical and Investigational Science Institute (CTSI) at USF.

Study Procedure - Those selected will be required to travel to the study site a total of 3 times for 2 days each at their own expense (some assistance may be available through the Foundation for Angelman Syndrome Therapeutics, visit www.cureangelman.org). It is important that you seriously consider your ability to complete the study. The number of participants we are allowed to enroll is strictly governed and funding is limited. It is imperative data is collected from each of the 24 participants to ensure the best possible results. We do not know if your child will benefit from receiving this medication, which is why we are doing this study.

During the visits your child will be asked to provide a blood sample and undergo an electroencephalogram gram (EEG), physical examination as well as behavioral assessments. During the first visit, the study drug, minocycline, will be dispensed to you. You will be asked to administer the study drug to your child twice daily. You will also be asked to log the administration to confirm compliance with the study regimen. A telephone interview will be conducted with you after 4 weeks of treatment to assess drug tolerance and to record any changes you may have observed. The study medication will be discontinued after 8 weeks of treatment. At the same time point, you will have to return to the study site for a follow up visit identical to the primary visit. The final follow up visit will occur at the 16 week time point (8 weeks following the minocycline treatment). This visit will be identical to the first two visits and will assess the lasting effects of the medication. Below is a summary of the study procedures.

Summary of Study Procedures:

1. Recruitment Begins - Interested parents contact the study staff via the internet form.
2. Prescreening packets are sent - Informed Consent Document, Health Information Release & Primary Care Physician (PCP) questionnaire
3. Eligibility Determined for 30 potential participants
4. Random Selection of 24 participants
5. Baseline Testing - Informed Consent Obtained, Lab work and EEG performed History and Physical exam performed
6. Enrollment - Study Neurologist confirms the participant meets the study criteria.
7. Behavioral Assessment
8. Minocycline Administration
9. Telephone Interview (4 weeks)
10. Discontinue Minocycline (8 weeks)
11. Follow up Assessment (8 weeks)
12. Telephone Interview (12 weeks)
13. Final Follow up assessment (16 weeks)

At the bottom of the page you will find a link to the weeberlab.com/clinical_trials.html website. There you will be able to submit your contact information.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is between the ages of 4 to 12 years old.
2. The participant has been previously diagnosed with AS by clinical evaluation.
3. The participant's diagnosis has molecular confirmation (e.g. karyotyping, fluorescent in situ hybridization (FISH), DNA methylation test or sequencing of the ubiquitin-protein ligase E3A gene) of the diagnosis.
4. The participant has a CGI-Severity Score of at least 4 indicating a moderate level of behavioral difficulty.
5. The participant is male or female.
6. The participant has an acceptable surrogate capable of giving consent on the participant's behalf.

Exclusion Criteria:

1. The participant was diagnosed with AS with no identifiable molecular abnormality.
2. The participant has a known allergy to MC or tetracycline.
3. The participant is currently enrolled in a study in which a drug, vitamin or dietary manipulation is used in the treatment of AS.
4. The participant suffers from severe or uncontrolled seizures or any other medical condition rendering the patient unstable.
5. The participant suffers from cardiovascular, respiratory, liver, kidney or hematologic disease.
6. The participant suffers from liver disease or elevated liver function tests.
7. The participant has a history of neutropenia, anemia or thrombocytopenia.
8. The participant has a history of systemic lupus erythematosus or an anti-nuclear antibody (ANA) titer or >1:40.
9. The participant is pregnant or at risk of becoming pregnant (sexually active females).
10. The participant experiences persistent psychotic symptoms.
11. The participant (or a parent/caregiver) is not willing to participate in clinic visits.
12. The participant experiences severe symptoms judged to likely to endanger the participant's safety or the safety of others.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin J Weeber, Ph.D., Principal Investigator — University of South Florida
Locations (1):
- Univeristy of South Florida, Tampa, Florida, United States

REFERENCES:
- [Derived] Grieco JC, Ciarlone SL, Gieron-Korthals M, Schoenberg MR, Smith AG, Philpot RM, Heussler HS, Banko JL, Weeber EJ. An open-label pilot trial of minocycline in children as a treatment for Angelman syndrome. BMC Neurol. 2014 Dec 10;14:232. doi: 10.1186/s12883-014-0232-x. PMID 25491305
- See also: If your interested in participating, click this link and submit your contact information. — http://weeberlab.com/clinical_trials.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Children With Angelman Syndrome
Started | 25
Completed | 24
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Children With Angelman Syndrome
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.6 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Bayley Scales of Infant and Toddler Development, 2nd Edition (BSID-II) Score at Baseline, 8 Weeks After Treatment, and at 16 Week Follow-up
Description: The primary outcome measure consists of improvement in raw and standard scores on the Bayley Scales of Infant and Toddler Development when post Minocycline administration results are compared to baseline results. This is an individually administered test used to asses developmental functioning. The Bayley scales are typically used for ages 1-42 months, and can be utilized to identify developmental delay by evaluating five major areas of development: cognitive, communication, physical, social/emotional, and adaptive.
  The score ranges for each subscale are as follows: Cognitive, 0-91; Communication, 0-75; Receptive Language, 0-49; Expressive Language, 0-48; Gross Motor, 0-72; Fine Motor, 0-66; Self-Care, 0-72; and Self-Direction, 0-75.
  Fine and Gross Motor scores were summed for the Motor domain; Receptive and Expressive Language were combined for the Language domain.
  Increase in raw score indicates improvement in the specific subdomain for each of the listed scales.
Time Frame: Baseline, 8 weeks & 16 weeks
Measure: Mean (Standard Deviation); unit: Scores on Scale
Arm/Group | Baseline Measures | 8 Weeks After Treatment With Minocycline | 16 Weeks-After 8 Week Washout
Number analyzed (Participants) | 24 | 24 | 24
Scores on Scale
  Cognitive | 26.4 (2.48) | 31.7 (1.83) | 30.7 (2.09)
  Communication | 18.9 (1.6) | 22.8 (1.69) | 23.5 (1.88)
  Receptive Language | 13.4 (0.61) | 13.7 (0.81) | 13.8 (0.68)
  Expressive Language | 10.1 (0.76) | 11.8 (0.75) | 11.2 (0.68)
  Gross Motor | 41.3 (1.69) | 40.5 (1.6) | 42.8 (1.12)
  Fine Motor | 19.4 (1.05) | 19.8 (1.47) | 22.4 (1.5)
  Self-Care | 37.8 (1.81) | 40.6 (1.84) | 40 (1.99)
  Self-Direction | 3.8 (2.24) | 38.1 (1.98) | 39.5 (1.94)

2. Secondary Outcome: Normalization of the EEG (Electroencephalogram) Signature
Description: A scoring system was used to evaluate several aspects of the EEG recordings regardless of whether or not they were a part of AS specific EEG patterns. Points were assigned when a particular characteristic was observed. For instance, when evaluating the EEG background, 1 point was assigned if primarily theta waves (mild slowing, >50%) were observed. When a mixture of theta and delta waves (moderate slowing) were observed, 2 points were assigned. When primarily delta waves (severe slowing, >50%) were recorded 3 points were assigned. Other EEG characteristics were also examined including occipital rhythm (normal-1, slow-2 and absent-3), rhythmic theta (present <50% of time-1, present >50% of time-2) rhythmic delta (present-3) and epileptiform abnormalities (present-1, focal-1, multifocal-1, generalized-1, seizure-2). The points were totaled resulting in a total score, ranging from 0 (most normal) to 24 (most abnormal).
Time Frame: Baseline, 8 and 16 weeks
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Baseline Measures | 8 Weeks After Treatment With Minocycline | 16 Weeks-After 8 Week Washout
Number analyzed (Participants) | 24 | 24 | 24
Score | 9.16 (3.47) | 8.76 (2.8) | 8.17 (3.47)

3. Secondary Outcome: Vineland Adaptive Behavior Scale, 4th Edition (Vineland-II)Score at Baseline, 8 Weeks After Treatment, and at 16 Week Follow-up
Description: This test is to measure the adaptive behaviors; the ability to adapt to changes in one's environment, learn new everyday skills and level of independence. It measures social and personal skills via five major domains: communication, daily living skills, socialization, motor skills, and a maladaptive behavioral index. These scales can be used to support the diagnosis of intellectual and developmental disability.
  The score ranges for each subdomain are as follows: Receptive Communication, 0-108; Expressive Communication, 0-308; Fine Motor, 0-196; Gross Motor, 0-228; Personal Daily Living Skills, 0-268; Domestic Daily Living Skills, 0-184; Community Daily Living Skills, 0-348; Internalizing Maladaptive Behavior, 0-22; and Externalizing Maladaptive Behavior, 0-20. These raw scores are allocated into the five major domains, and standardized for analysis of results.Increase in raw score indicates improvement in the specific subdomain for each, except for Maladaptive Behavior Scales.
Time Frame: Baseline, 8 and 16 weeks
Measure: Mean (Standard Deviation); unit: Scores on Scale
Arm/Group | Baseline Measures | 8 Weeks After Treatment With Minocycline | 16 Weeks-After 8 Week Washout
Number analyzed (Participants) | 24 | 24 | 24
Scores on Scale
  Receptive Communication | 30.28 (8.10) | 36.4 (12.08) | 33.88 (11.00)
  Expressive Communication | 41.84 (15.11) | 44.28 (14.95) | 43.79 (12.64)
  Fine Motor Ability | 98.96 (35.60) | 101.2 (39.62) | 95.38 (38.45)
  Gross Motor Ability | 48.28 (16.62) | 48.92 (16.62) | 49.38 (15.90)
  Daily Living Skills - Personal | 53.8 (28.05) | 59.12 (28.73) | 56.38 (24.28)
  Daily Living Skills - Domestic | 2.6 (4.76) | 3.84 (7.46) | 2.67 (4.49)
  Daily Living Skills - Community | 6.04 (9.09) | 7.44 (9.57) | 7.08 (7.92)
  Maladaptive Behavior - Internalizing | 6.68 (2.23) | 5.48 (2.35) | 5.71 (2.54)
  Maladaptive Behavior - Externalizing | 5.64 (2.87) | 4.68 (2.87) | 6.00 (6.12)

4. Secondary Outcome: Preschool Language Scale, Fourth Edition (PLS-4)Score at Baseline, 8 Weeks After Treatment, and at 16 Week Follow-up
Description: This test is used to evaluate the development of expressive and receptive language development. It also can be used to assess behaviors considered to be language precursors. The PLS use a play-based assessment to provide a comprehensive developmental language appraisal. These scales assess auditory and expressive comprehension. The score ranges for the two subdomains of this measure depend on 16 chronological age ranges from birth - 7 years, with a score range of 0-62 in Auditory Comprehension and 0-68 for Expressive Communication in a 7 year old. Minimum range: 50 (lower language abilities) Maximum range: 150 (higher language abilities). The PLS use a play-based assessment to provide a comprehensive developmental language appraisal. Increase in raw score indicates improvement in the specific subdomain. These raw scores are standardized for analysis and comparison. Standardization does not impact the interpretation of the results
Time Frame: Baseline, 8 and 16 weeks
Measure: Mean (Standard Deviation); unit: Scores on Scale
Arm/Group | Baseline Measures | 8 Weeks After Treatment With Minocycline | 16 Weeks-After 8 Week Washout
Number analyzed (Participants) | 24 | 24 | 24
Scores on Scale
  Auditory Comprehension | 17.664 (3.43) | 18.25 (2.86) | 20.47 (3.42)
  Expressive Communication | 16.28 (5.72) | 16.63 (4.62) | 17.48 (4.69)
  Total Language Ability | 34.20 (7.87) | 34.88 (6.65) | 38.83 (6.43)

5. Secondary Outcome: Clinical Global Impressions Severity Scale Score at Baseline, 8 Weeks After Treatment, and at 16 Week Follow-up
Description: The CGI is a brief assessment used by the clinician to describe the participants condition before and after the administration of a study medication.It is a research rating tool that physicians use to provide a timely assessment of a clinician's view of a particular patient's global functioning before and after the usage of a study medication. The CGI is used to measure the change since the initiation of treatment; both measures 10 questions on a seven-point Likert-type scale ranging from ranging from 1 to 7 points, equaling 10-70 points total, from which the mean is attained. A decrease in mean score indicates improvement in the specific sub-domain.
Time Frame: Baseline, 8 & 16 weeks
Measure: Mean (Standard Deviation); unit: Scores on Scale
Arm/Group | Baseline Measures | 8 Weeks After Treatment With Minocycline | 16 Weeks-After 8 Week Washout
Number analyzed (Participants) | 24 | 24 | 24
Scores on Scale | 5.5 (1.1) | 4.88 (1.03) | 5.08 (1.25)

ADVERSE EVENTS:
Time Frame: Events were reported to the investigator by the parents of participant throughout the 16 week trial.
Arm/Group | Children With Angelman Syndrome Receiving Minocycline
Serious Adverse Events (participants affected / at risk) | 3/25
Other Adverse Events (participants affected / at risk) | 9/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Children With Angelman Syndrome Receiving Minocycline (N=25)
Seizure (Congenital, familial and genetic disorders) | 3 — Seizure is a common characteristic of Angelman Syndrome (80%). Parent reported occurrence of seizure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Children With Angelman Syndrome Receiving Minocycline (N=25)
Lethargy/Sleepiness (Congenital, familial and genetic disorders) | 2
Difficulty Ambulating (Congenital, familial and genetic disorders) | 2
Darkening/discoloration over the anterior tibia (Congenital, familial and genetic disorders) | 1
Commencement of Menstruation (Congenital, familial and genetic disorders) | 1
Urinary Tract Infection (Congenital, familial and genetic disorders) | 1
Influenza Type A (Congenital, familial and genetic disorders) | 1
Feminine yeast Infection (Congenital, familial and genetic disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No